CLINICAL TRIAL: NCT05780840
Title: Protection Against Visible Light by Dihydroxyacetone in Erythropoietic Protoporphyria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ida M. Heerfordt, Principal Investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dihydroxyacetone
Record Dates: First submitted 2023-02-22; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Erythropoietic Protoporphyria
Keywords: Dihydroxyaceton; Erythropoietic protoporphyria; Light protection; Protoporphyrin IX; Self-tanning; Skin
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — Dihydroxyacetone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dihydroxyacetone (Experimental)
  Interventions: Other: Dihydroxyacetone; Other: Placebo
- Placebo (Placebo Comparator)
  Interventions: Other: Dihydroxyacetone; Other: Placebo

INTERVENTIONS:
Other: Dihydroxyacetone — Application of 10% dihydroxyacetone (2 mg per square cm skin)
Other: Placebo — Application of lotion to the skin (2 mg per square cm skin)

SUMMARY:
What is the visible light protective effect of dihydroxyacetone in individuals with erythropoietic protoporphyria? This will be tested in this randomized blinded placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with erythropoietic protoporphyria
* At least 18 years of age
* Obtainment of written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Use of dihydroxyacetone at the treatment or placebo fields within the last two week
* Sun exposure of the treatment or placebo fields within the last two week
* Use of suncreen or other local treatment on the treatment or placebo fields during the study period (two days)
* Allergy to adhesive bandages, dihydroxyacetone or lotion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Visible light exposure dose to onset of first skin symptom | Meassurement one day after dihydroxyacetone application
  Assessed by phototesting

SECONDARY OUTCOMES:
Change in skin color from before treatment to one day after treatment | Meassurement of skin color just before dihydroxyacetone application and one day after application.
  Assessed by color scale. The color scale is presented in DOI: 10.1111/phpp.12458.
  It is a seven-point scale to assess skin color from light to dark. We expect that a large change in skin color will give the best effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Ida Marie Heerfordt, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Study protocol — https://doi.org/10.1016/j.pdpdt.2023.103302